CLINICAL TRIAL: NCT02096887
Title: Effect of Patient Awareness and Education on Compliance and Cardiovascular Risk Factor Control
Brief Title: Effect of Patient Education on Compliance and Cardiovascular Risk Parameters
Acronym: FAILAKA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kuwait Institute for Medical Specialization (Other Government)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Dr. Samia Almusallam, Director of the family medicine residency program, Kuwait Institute for Medical Specialization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WS964765
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Cardiovascular Risk Factors
Keywords: education; compliance; risk factors
MeSH Terms: conditions — Patient Compliance | interventions — Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient Education (Other): Patient Education
  Interventions: Behavioral: Patient Education

INTERVENTIONS:
Behavioral: Patient Education — Patient Education using the following two instruments:
  1. Framingham Risk Score calculator:
  2. Know your numbers patient booklet

SUMMARY:
Patient's awareness of their risk factors for heart disease and their active involvement in their own management plan can help improve their adherence to treatment and their risk profile. The purpose of this study is to investigate the influence of patient education and awareness of heart disease risk factors on compliance to medication and lifestyle modification.

DETAILED DESCRIPTION:
Prospective cluster randomized interventional study with primary health care clinics as clusters.Clinics will be randomized to conventional care or to structured patient education in addition to care. Trained physicians will extract information from the patient medical record and will conduct a personal interview with the participants, after they finish with their routine visit, to fill a case report form (CRF)

CRF will include the following items:

* Patient Demographics,
* Socioeconomic: income, employment and education
* Past Medical History
* Smoking history
* Alcohol use
* Medications
* Adherence: Morisky scale
* Examination: BP, weight, height, waist
* Investigations: LDL-C, HbA1C 2.Compliance/adherence to the medication will be measured by using the Morisky scale, which is a validated scale for measuring adherence in hypertension and diabetic patients among other disease.

Patients attending clinics that are randomized to structured patient education will receive education targeting all the risk factors they have. They will be informed about specific evidence -based target values they should achieve for each of the risk factors. Their compliance to prescribed medications will be encouraged and specific advice about improving compliance will be given. To achieve this physicians in the education clinics are going to use two items:

1. Framingham Risk Score calculator.
2. Know your numbers patient booklet.

Follow up visits will be scheduled at 2 months, 6 months and 12 months after the initial visit. For patients in both education and conventional clinics, compliance to medications will be assessed and the degree of risk factor control will also be determined through specific measurements that include number of cigarettes smoked, systolic and diastolic blood pressure, body mass index and waist circumference, HBA1C and LDL values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one or more CVD risk factors will be consecutively enrolled, smokers and obese patients should have an additional risk factors
* The risk factors are based on Framingham Risk Score calculator and include smoking, high blood pressure, high blood cholesterol ,diabetes and being overweight or obese
* All participants must be adults (30 -70 years of age) who give an informed consent
* All participants should be of Kuwaity nationality, literate and fluent in either Arabic or English
* Patients are likely to be available for a one year follow up

Exclusion Criteria:

* Patients with mental disability or severe psychiatric disorder who are unable to provide informed consent or participate in educational activities.
* Patients with severe visual or hearing disability that will prevent participation in the educational activity
* Patients <30 years or >70 years of age
* Illiterate patients
* Non Kuwaity nationals
* Patients who are not permanently resident in Kuwait
* Patient who refuse to provide the informed consent

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
cardiovascualr risk factor control | 12 months
  Cardiovascular risk factors control as assessed by the following parameters: HbA1C, Blood pressure, LDL-C, BMI and smoking cessation
medication compliance | 12 months
  Medication compliance as assessed by Morisky scale

CONTACTS AND LOCATIONS:
Overall Officials: Samia Almusallam, FRCGP, Principal Investigator — Kuwait Institute for Medical Specialization; Maleka M Serour, MRCGP/ INT, Principal Investigator — Kuwait Institute for Medical Specialization; Wafa A Rashed, FRCP, Principal Investigator — Ministry of Health -Mubarak Hospital- Cardiology unit